CLINICAL TRIAL: NCT06477042
Title: Act on Quality of Life in Poor Prognosis Aortic Stenosis Patients
Brief Title: Act on Quality of Life in Patients With aortIc Stenosis
Acronym: ALPINIST
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0930
Record Dates: First submitted 2024-06-18; First posted 2024-06-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Severe Aortic Stenosis
Keywords: TAVI; quality of life; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Poor prognosis patients: Patients will performed the Quality Of Life Questionnaire (EQ-5D-5L) and the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) at baseline (day of the TAVI procedure) and 2 months post-TAVI. The CAPRI score will be calculated from the data of the pre TAVI assessment at the end of study participation (12 months) and will determine the group of the patient. The higher the score, the worse the prognosis.
  Interventions: Other: Kansas City Cardiomyopathy Questionnaire (KCCQ-12) score
- Intermediate prognosis patients: Patients will performed the Quality Of Life Questionnaire (EQ-5D-5L) and the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) at baseline (day of the TAVI procedure) and 2 months post-TAVI. The CAPRI score will be calculated from the data of the pre TAVI assessment at the end of study participation (12 months) and will determine the group of the patient. The higher the score, the worse the prognosis
  Interventions: Other: Kansas City Cardiomyopathy Questionnaire (KCCQ-12) score

INTERVENTIONS:
Other: Kansas City Cardiomyopathy Questionnaire (KCCQ-12) score — Change in quality-of-life score assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) between the 2-month early visit and inclusion in the poor-prognosis group.

SUMMARY:
Aortic stenosis (AS) is a degenerative process affecting the aortic valve that leads to sclerosis of the valve and limits its opening during cardiac contractions. The prognosis is poorly, with survival rates of only 15-50% at 5 years. AS has a major impact on quality of life, with severely limiting symptoms (dyspnea, chest pain,…) often leading to repeated hospitalizations. It is the most common valvular disease in Europe and North America, and its prevalence is increasing as the population ages. In Europe, 17% of the population is aged 65 or over; in France, this proportion will reach 30% by 2030, corresponding to 16 million people. The incidence of aortic valve sclerosis (early stage AS) is around 25% at age 65, rising to 48% after age 75. The prevalence of aortic valve disease is likely to continue to rise, given the expected evolution of the age pyramid.

There is no medical treatment able to slow down the degenerative process of the valve, and the only treatment is aortic valve replacement when the AS becomes constricted and the patient is eligible for an intervention. Aortic valve replacement has historically been performed surgically, with open-chest surgery to remove the damaged valve and replace it with a mechanical or biological valve prosthesis. Now Transcatheter Aortic Valve Implantation (TAVI) has replaced this procedure. This involves inserting a bioprosthesis crimped into a stent via an endovascular route, i.e. without opening the thorax. Deployment of the stent crushes the native valve, leaving the functional bioprosthesis in place.

Initially developed for patients contraindicated to surgery, TAVI is now offered as a first-line treatment for patients aged 75 and over.

Inexistent before 2010, the number of TAVIs equalled the number of surgeries by 2015, and TAVIs currently account for ¾ of aortic valve procedures (unpublished data).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic aortic stenosis (exertional dyspnea, angina, malaise/syncope)

  * Indication for TAVI (valve area 1 cm² or 1 cm²/m² body surface area or mean transvalvular aortic gradient > 40 mmHg on ultrasound) validated in Heart Team
  * Charlson score ≥ 5
  * Social health care insurance affiliation

Exclusion Criteria:

* Patient refusing TAVI procedure
* CT scan not performed during the pre-TAVI assessment
* Patient unable to understand or answer quality-of-life questionnaires
* Pregnant or breast-feeding women
* Patients participating in other interventional research that may interfere with the present study with an exclusion period still in progress
* Persons under judicial protection
* Patients under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with indication of TAVI followed in four french cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-12-19 (Estimated); Study Completion 2027-12-19 (Estimated)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) score variation between the 2-months visit and inclusion. | Day 0 and Month 2
  Change in quality-of-life score assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) between the 2-month early visit and inclusion in the poor-prognosis group. The KCCQ-12 contains four subdomains: Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Cardiologie - CHU Clermont Ferrand, Clermont-Ferrand
  - Service de Cardiologie, Lille
  - Service de Cardiologie, Lyon
  - Service de Cardiologie - Institut Thorax Nantes, Nantes